CLINICAL TRIAL: NCT01416454
Title: Thromboelastography to Assess Age-Related Coagulation Differences in Patients Undergoing Elective Cesarean Delivery.
Brief Title: Thromboelastography to Assess Age-Related Coagulation Differences in Patients Undergoing Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SU-11192010-7216; 19878 (Registry Identifier: Stanford University)
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Thrombophilia
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elective Cesarean delivery, age <35 yrs: Women undergoing elective cesarean delivery with a spinal anesthetic who are less than 35 y of age (at the time of delivery).
- Elective Cesarean delivery, age =>35 yrs: Women undergoing elective Cesarean delivery with a spinal anesthetic who are => 35 yrs of age (at the time of delivery).

SUMMARY:
The purpose of the study is to assess potential age-related differences on coagulation profile of patients undergoing Cesarean Section, using thromboelastography (TEG). The investigators will compare coagulation data collected from the study to assess potential differences in coagulation parameters for the following age groups: (i) women less than 35 yrs (ii) women 35 yrs or older.

DETAILED DESCRIPTION:
The purpose of the study is to assess potential age-related differences on coagulation profile of patients undergoing Cesarean Section, using thromboelastography (TEG). The investigators will compare coagulation data collected from the study to assess potential differences in coagulation parameters for the following age groups: (i) women less than 35 yrs (ii) women 35 yrs or older. This study will allow us to collect more information about differences regarding coagulation profile in patients undergoing cesarean section who are less than 35 y vs. 35y or older. This information will add to current knowledge base about potential risk for thrombotic events according with age.

All obstetric patients presenting for elective Cesarean delivery (CD) will be informed about the study prior to and on admission to the labor and delivery unit. Patients will be informed at parents' education classes (during education sessions by obstetric anesthesiologists who are also members of the research team). Potential participants will be approached by a member of the research team prior to surgery. A study investigator will obtain patient written informed consent.

Pre-operatively, blood sampling will take place by venepuncture for the following analysis:

Hematocrit, Platelet count (which are part of standard of care), TEG, prothrombin time (PT), Partial Thromboplastin Time (PTT), International Normalized Ratio (INR), fibrinogen (for research purposes only, unless they are needed for clinical purposes).

The investigators would prefer to avoid taking blood samples from indwelling peripheral IV lines, as the samples will likely be diluted with intravenous fluid and therefore may significantly affect blood sampling analysis. The volumes of blood necessary for TEG analysis are extremely small (1 ml - less than half of a teaspoon - per TEG analysis; total =3 samples), and therefore will not significantly affect any potential degree of hemorrhage or total blood loss incurred. The volumes of blood for laboratory analysis will also be small (4-5 ml - about 1 teaspoon - for each research sample: total =3 samples), and will not affect overall blood loss. No randomization will be possible. TEG and laboratory samples will be taken at the following time intervals: prior to anesthesia in the preoperative holding unit, post-operative days one and three.

Data will be assessed for normality using normality plots and the Kolmogorov-Smirnov test. Normally and non-normally distributed TEG parameters before and after CD (PACU samples) will be assessed by using the paired t-test and Wilcoxon signed-rank test respectively. The percentage change from baseline for each TEG parameter and Hb before and after CD will also be calculated. Longitudinal analysis of individual changes for each TEG parameter will be performed using mixed effects regression modeling, due to the non-uniformity of time-intervals and to account for correlation among repeated measurements on the same participants. The investigators will examine longitudinal models for individual TEG parameters as a dependent measure, with study group as a fixed factor, and number of previous cesarean section, total blood loss, IV fluids, platelet count and fibrinogen counts as potential covariates (tbc). Separate models will incorporate age as continuous independent variable (as both a fixed and random effect). The investigators will analyze these data using SAS version 9.2 (SAS Institute, Cary, N.C., USA).

Study data will be stored in secured, locked storage boxes which will only be accessed by study investigators. Samples and labels will be identified using a numerical system based allocated prior to the start of the study. Only investigators directly involved in the study will have access to the study data and other related documents.

Study data will be protected as follows:

Hard data will be stored in secure box-files kept in locked file cabinets; databases with study data will be password-protected. Study information will be coded in advance using a numerical coding system not linked to the patients' medical record number or other PHI. Coding will be performed when data is entered into the database. Only study investigators will have access to the coding system for de-identifying data. All codes used to protect study data and confidential information will be used solely by study investigators. All codes used for data- protection will be known only to the study investigators, and software-protection and encryption programs will be used as appropriate.

TEG will be performed by study investigators on the labor and delivery unit. Blood samples will be destroyed after TEG analysis. Other laboratory samples will be analyzed as per normal procedure.

Electronic data will be stored at the Stanford File Management Tool. Only researchers and research staff will be granted password-protected access to identifiable and coded data stored on this server.

All persons involved in this study will receive appropriate training and abide by confidentiality guidelines to protect the subject's privacy. All HIPAA rules and regulations will be strictly followed.

ELIGIBILITY:
Inclusion Criteria:

* All obstetric patients with singleton pregnancies admitted to the labor and delivery unit at LPCH who undergo elective Cesarean delivery with neuraxial anesthesia.
* We will enroll only healthy patients with singleton pregnancies and whose pregnancy is not result of in vitro fertilization.

Exclusion Criteria:

* Patients with underlying coagulation disorders.
* Patients with thrombocytopenia.
* Patients with pregnancy-induced hypertension, pre-eclampsia.
* Patients requiring the following medications prior to surgery: non-steroidal anti-inflammatories, aspirin, anticoagulants.
* Patients requiring non-elective Cesarean delivery.
* Patients with significant obstetric or medical disease.
* No patients <18 years of age will be recruited.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study population will be obstetric patients undergoing delivery on the labor and delivery unit at Lucile Packard Children's Hospital (LPCH).
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Thromboelastography parameters | 3 days
  Thromboelastography parameters include:
  Reaction (r) time Clot Formation (k) time Alpha Angle Maximum Amplitude (MA) Time to maximum rate of thrombus generation (Tmax) Maximum rate of thrombus generation (MRTG) Total Thrombus generated (TTG)

SECONDARY OUTCOMES:
laboratory coagulation parameters | 3 days
  * Prothrombin time
  * Activated partial thromboplastin time
  * Fibrinogen level.

CONTACTS AND LOCATIONS:
Overall Officials: Alex James Butwick, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] James AH. Venous thromboembolism in pregnancy. Arterioscler Thromb Vasc Biol. 2009 Mar;29(3):326-31. doi: 10.1161/ATVBAHA.109.184127. PMID 19228606
- [Background] Bates SM, Greer IA, Pabinger I, Sofaer S, Hirsh J. Venous thromboembolism, thrombophilia, antithrombotic therapy, and pregnancy: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):844S-886S. doi: 10.1378/chest.08-0761. PMID 18574280
- [Background] Morris JM, Algert CS, Roberts CL. Incidence and risk factors for pulmonary embolism in the postpartum period. J Thromb Haemost. 2010 May;8(5):998-1003. doi: 10.1111/j.1538-7836.2010.03794.x. Epub 2010 Feb 1. PMID 20128859
- [Background] Sharma SK, Philip J, Wiley J. Thromboelastographic changes in healthy parturients and postpartum women. Anesth Analg. 1997 Jul;85(1):94-8. doi: 10.1097/00000539-199707000-00017. PMID 9212129
- [Background] Saha P, Stott D, Atalla R. Haemostatic changes in the puerperium '6 weeks postpartum' (HIP Study) - implication for maternal thromboembolism. BJOG. 2009 Nov;116(12):1602-12. doi: 10.1111/j.1471-0528.2009.02295.x. Epub 2009 Aug 14. PMID 19681851
- [Background] Ng KF. Changes in thrombelastograph variables associated with aging. Anesth Analg. 2004 Aug;99(2):449-54, table of contents. doi: 10.1213/01.ANE.0000133140.75831.1E. PMID 15271723
- [Derived] Butwick A, Gutierrez MC, Hilton G. The impact of advanced maternal age on peripartum thromboelastographic coagulation profiles: a prospective observational exploratory study. Can J Anaesth. 2015 May;62(5):504-12. doi: 10.1007/s12630-014-0300-0. Epub 2014 Dec 31. PMID 25549988